CLINICAL TRIAL: NCT01433484
Title: Community-Based Lifestyle Intervention to Reduce CVD Risk & Disparities in Risk
Brief Title: Heart-Healthy Lenoir Lifestyle Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-0395LS; P50HL105184 (NIH)
Record Dates: First submitted 2011-08-30; First posted 2011-09-14 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2015-08

CONDITIONS: Cardiovascular Disease; Obesity
Keywords: cardiovascular disease; coronary heart disease; obesity; weight loss; genomics
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Coronary Disease; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance of Weight Loss--Control (Active Comparator): The control arm will receive bi-monthly telephone contacts during the one-year maintenance phase.
  Interventions: Behavioral: Maintenance of Weight Loss--Control
- Maintenance of Weight Loss--Experimental (Experimental): The experimental arm will receive monthly telephone contacts for one year during the maintenance phase.
  Interventions: Behavioral: Maintenance of Weight Loss--Experimental

INTERVENTIONS:
Behavioral: Maintenance of Weight Loss--Control — As the maintenance of weight loss randomized trial does not begin until a year after the start of this study, the intervention and control conditions are not yet specified. This will occur before randomization and this section will be updated before the first participant is randomized.
  Arms: Maintenance of Weight Loss--Control
Behavioral: Maintenance of Weight Loss--Experimental
  Arms: Maintenance of Weight Loss--Experimental

SUMMARY:
This study aims to reduce cardiovascular disease (CVD) risk and disparities in risk by improving lifestyle factors which underlie the development of CVD. The first steps will involve conducting a comprehensive formative evaluation to assess individual, interpersonal, organizational, community, and policy factors relevant to CVD risk and risk reduction in Lenoir County. This will be followed by a community-based lifestyle intervention program designed to improve eating patterns, promote physical activity, and for those who are interested, support weight loss. A randomized trial comparing the effectiveness of two community based weight maintenance interventions will also be conducted. Community-wide policy and environmental change interventions will also be implemented to support the individual-level interventions, including partnerships with businesses to promote a healthy environment through innovative economic opportunities. In addition, this project will explore genetic factors associated with cardiovascular disease risk and treatment success.

DETAILED DESCRIPTION:
The lifestyle intervention will enroll 350 participants. The initial lifestyle component of this study, which lasts for 4-6 months, will be provided to all participants. Participants may chose from one of two intervention formats, each with 4 contacts: individual counseling with at least one face-to-face visit and the rest face-to-face or by phone or 4 group sessions. The dietary intervention will focus on improving fat and carbohydrate quality. For fat intake, the goals include 2-4 servings per day of polyunsaturated fat primarily from plant sources and minimal intake of trans fat. For carbohydrate intake, the goals include increased intake of whole grains, fruits and vegetables, and beans and reduced consumption of refined carbohydrates. The physical activity intervention will primarily focus on walking with a goal of 7500 to 10,000 steps per day or, for those who do not wish to use a pedometer, 30 minutes of walking a day. Muscle strengthening activities will also be recommended. At the 4-6 month follow-up measures, those who wish to take part in a weight loss study may do so and those who do not will continue in a maintenance of lifestyle intervention.

The investigators anticipate approximately 200 participants will take part in the weight loss component of this study, which consists of a 6 month intensive weight loss intervention. Participants may choose from two intervention formats: 16 weekly group sessions or 5 group sessions and 10 phone counseling sessions. The weight loss goal will be 5% of body weight. At the conclusion of this program, those who lose at least 8 pounds and are willing to take part in a 1 year maintenance of weight loss intervention will be RANDOMIZED to one of two maintenance of weight loss programs. One maintenance arm will receive monthly telephone contacts for one year, while the other arm will receive bi-monthly phone contacts.

Follow-up measures for all participants will be at approximately 6, 12, 18, and 24 months.

Another related part of the project will use a systems approach to develop models integrating clinical and genomic data. Researchers have developed and tested an approach referred to as the SAMARA (Supporting A Multidisciplinary Approach to Research in Atherosclerosis) Project that applies recent, major advances in biomedical and computational sciences at UNC to develop a deeper understanding of human CVD. The Heart-Healthy Lenoir Project will expand studies into the community, using this methodology to: 1) determine the prevalence of genomic risk signatures in high-risk community populations using genome-wide Single Nucleotide Polymorphism (SNP) analysis; 2) develop novel genomic models incorporating high-risk features in this population; and 3) determine whether genomic signatures can be used to predict responsiveness to interventions that underlie CVD disparities. Participants who consent to this component of the project will have a blood specimen obtained at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. live in Lenoir County or a neighboring county in Eastern North Carolina
3. anyone enrolled in the Lifestyle study is eligible to participate in the genomics component of the project.

Exclusion Criteria:

1. non-English speaking
2. treatment of psychosis
3. alcohol or substance abuse within the two last years
4. history of malignancy, other than non-melanoma skin cancer, unless surgically cured > 5 years ago or in remission/well treated and not likely to have a negative effect on the patient's health over the next 2 years
5. estimated creatinine clearance less than 30 ml/min
6. lack of access to phone
7. advanced dementia
8. participants who have been diagnosed with a myocardial infarction within the past three months will be excluded from the study if they are unable to obtain written medical clearance from their clinician to participate in the study

Additional Exclusion Criteria - Weight Loss Intervention:

1. the investigators will not invite pregnant women to take part in the weight loss study.
2. if a woman becomes pregnant while taking part in this part of the study, we will withdraw her from the weight loss study and invite her to continue in the lifestyle study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Cohort study: fruit and vegetable intake at 6 months | 6 months
  Fruit and vegetable intake will be measured by the Block fruit and vegetable sceener and by blood carotenoids
Embedded randomized trial: maintenance of weight loss | 1 year after maintenance of weight loss trial begins
  Weight will be measured by electronic scale

SECONDARY OUTCOMES:
Physical activity | 6m, 12m, 18m, 24 m
  Measured by questionnaire and pedometer
Blood pressure | 6, 12, 18, 24 months
  measured by automated device
Blood lipids | 12, 24 months
  total and HDL cholesterol measured by commercial lab
A1c | 6, 12, 24 months
  measured by commercial lab
Fruit and vegetable intake at 6 months | 12, 18, and 24 months
  Measured by Block fruit and vegetable screener
Weight | 6, 12, 18, 24
  Measured by electronic scale
Health related quality of life | 6, 12, 24 months
  SF-12 instrument
Genomic predictors of lifestyle change | 6-, 12-, 18- and 24-month follow-up
  A systems approach to developing genomic models integrating clinical and genomic data.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Keyserling, MD, MPH, Principal Investigator — UNC-Chapel Hill
Locations (1):
- Heart Healthy Lenoir Project, Kinston Enterprise Center, Kinston, North Carolina, United States

REFERENCES:
- [Derived] Embree GG, Samuel-Hodge CD, Johnston LF, Garcia BA, Gizlice Z, Evenson KR, DeWalt DA, Ammerman AS, Keyserling TC. Successful long-term weight loss among participants with diabetes receiving an intervention promoting an adapted Mediterranean-style dietary pattern: the Heart Healthy Lenoir Project. BMJ Open Diabetes Res Care. 2017 Mar 29;5(1):e000339. doi: 10.1136/bmjdrc-2016-000339. eCollection 2017. PMID 28405344
- [Derived] Keyserling TC, Samuel-Hodge CD, Pitts SJ, Garcia BA, Johnston LF, Gizlice Z, Miller CL, Braxton DF, Evenson KR, Smith JC, Davis GB, Quenum EL, Elliott NT, Gross MD, Donahue KE, Halladay JR, Ammerman AS. A community-based lifestyle and weight loss intervention promoting a Mediterranean-style diet pattern evaluated in the stroke belt of North Carolina: the Heart Healthy Lenoir Project. BMC Public Health. 2016 Aug 5;16:732. doi: 10.1186/s12889-016-3370-9. PMID 27495295
- See also: Provides information about this study — http://www.hearthealthylenoir.com